CLINICAL TRIAL: NCT04795609
Title: Effect of a Post-operative Protocol of Early Mobilization on Functional Recovery and Postoperative Complications After Immediate Internal Pudendal Artery Perforator Flap Reconstruction for Irradiated Abdominoperineal Resection Defects: a Prospective, Randomized and Controlled Clinical Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP1561
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator): Early mobilization postoperative programme based on supervised aerobic exercise, resistance and flexibility training or to standard rehabilitation care
  Interventions: Other: Early mobilization strategy adapted after immediate internal pudendal artery perforator flap reconstruction for abdominoperineal resection (intervention group).
- Control group (No Intervention): Bed restriction strategy for 5 days

INTERVENTIONS:
Other: Early mobilization strategy adapted after immediate internal pudendal artery perforator flap reconstruction for abdominoperineal resection (intervention group). — Early mobilization strategy adapted after immediate internal pudendal artery perforator flap reconstruction for abdominoperineal resection (intervention group).
  1. Trunk control.
  2. Orthostatism.
  3. Walk training.
  4. Aerobic exercises.
  5. Muscle strengthening.
  Arms: Interventional group

SUMMARY:
Major abdominal oncology surgery is associated with substantial postoperative loss of functional capacity, and exercise may be an effective intervention to improve outcomes. The aim of this study was to assess efficacy, feasibility and safety of a supervised postoperative exercise programme in patients undergoing immediate internal pudendal artery perforator flap reconstruction for irradiated abdominoperineal resection defects.

We will perform a open label, parallel-arm, randomized trial in patients who underwent immediate internal pudendal artery perforator flap reconstruction for irradiated abdominoperineal resection defects in a tertiary university hospital.

Patients will be randomized to an early mobilization postoperative programme based on supervised aerobic exercise, resistance and flexibility training or to standard rehabilitation care - bed restriction for 5 days. The primary outcome will be inability to walk without human assistance at postoperative day 5 or hospital discharge.The secondary outcomes will be incidence of surgical complications, ability of walk assessed for the 6-minute walk test, incidence and intensity of fatigue measured by Piper's Revised Fatigue Scale, improvement of quality of life measured by EuroQuol-5D-5L Questionnaire, Incidence of deep venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing immediate internal pudendal artery perforator flap reconstruction for abdominoperineal resection .
2. Age ≥ 18 years.
3. Agreement to participate and signature of the informed consent form by the patient and / or family.

Exclusion Criteria:

1. Acute myocardial infarction (in the last 30 days) or Unstable angina.
2. Uncontrolled cardiac arrhythmia.
3. Symptomatic severe aortic stenosis or other symptomatic severe valve dysfunction.
4. Congestive heart failure NYHA III or IV.
5. Hemodynamic instability.
6. Venous thromboembolism.
7. Pericarditis, endocarditis or myocarditis.
8. Aortic dissection.
9. Septic shock.
10. Need for renal replacement therapy.
11. Thyrotoxicosis.
12. Presence of bone metastasis.
13. Osteomioarticular and neurological conditions that make it impossible to carry out the exercise program designed for this study.
14. Palliative procedures.
15. Inability to perform the exercises due to musculoskeletal or neurological changes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Capacity of functional walking. | 5 days.
  Capacity of functional walking, assessed by the patient's ability to cross the hospital room or the ability to walk 3 meters independently on the 5th postoperative day.

SECONDARY OUTCOMES:
Hospital stay. | 30 days.
  Hospital Stay.
Postoperative complications. | 30 days.
  Incidence of postoperative complications using the Clavien-Dindo classification.
Functional walking capacity, assessed by the 6-minute walk test. | 30 days.
  Functional walking capacity, assessed by the 6-minute walk test.
Incidence and intensity of fatigue measured by the Piper Revised Fatigue Scale. | 30 days.
  Incidence and intensity of fatigue measured by the Piper Revised Fatigue Scale.
Quality of life measured by the EuroQol-5D-5L Questionnaire. | 30 days.
  Quality of life measured by the EuroQol-5D-5L Questionnaire.
Incidence of deep venous thrombosis. | 30 days.
  Incidence of deep venous thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Caio Araujo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No